CLINICAL TRIAL: NCT03010722
Title: A Prospective Translational Study Investigating Molecular Predictors of Resistance and Response to Regorafenib Monotherapy in RAS Mutant Metastatic Colorectal Cancer
Brief Title: Prospective Translational Study Investigating Molecular Predictors of Resistance and Response to Regorafenib Monotherapy
Acronym: PROSPECT-R
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 4164
Record Dates: First submitted 2015-01-06; First posted 2017-01-05 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2017-01

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue and plasma samples will be retained for a maximum period of 20 years, according to UK regulatory approval policy and study protocol.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Regorafenib: 160 mg orally (po) od for 3 weeks of every 4-week cycle
  All patients will be required to have pre-treatment dynamic contrast enhance computed tomography (DECT) scan pre-treatment and at 8 weeks. Suitable patients will also be required to have dynamic contrast enhanced magnetic resonance imaging (DEC-MRI) and diffusion weighted (DW)-MRI, pre-treatment and at 2 weeks. All patients will also be required to have an Ultrasound (USS) or CT-guided biopsy of suitable metastatic lesion.
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — Patients meeting all of the inclusion criteria and none of the exclusion criteria will receive regorafenib 160 mg orally (po) od for 3 weeks of every 4-week cycle. Each cycle will comprise 3 weeks of treatment followed by 1 week without treatment, hereafter described as "3 weeks on/1 week off". Each 160-mg dose will include four regorafenib 40-mg tablets.
  Other Names: Stivarga

SUMMARY:
This is a single centre prospective biological translational research study involving the collection of tumour tissue, blood samples and clinical data from patients being treated with regorafenib for metastatic Colorectal Cancer (mCRC) at the Royal Marsden Hospital. Patients will be eligible for the study if they have a histological diagnosis of CRC, are refractory to standard available therapies with palliative intent for mCRC, have received prior treatment with at least one anti-VEGF antibody and chemotherapy drugs including fluorouracil (5FU) or capecitabine, oxaliplatin and irinotecan, and patients have RAS mutant tumours.

DETAILED DESCRIPTION:
This is an exploratory translational research study to obtain research biopsies of RAS mutant metastatic colorectal cancer (mCRC) tumour tissue prior to commencement of regorafenib multi-tyrosine kinase inhibitor (MKI) treatment targeting vascular endothelial growth factor receptor (VEGFR), tumour microenvironment and oncogenic driver alterations, and again at development of resistance. Candidate markers of resistance will be identified in tissue biopsies through genetic and other molecular analysis and parallel collection of serial blood specimens will facilitate the identification of resistance markers and the tracking of resistance evolution in circulating nucleic acids. Early dynamic contrast enhanced MRI (DCE-MRI) along with diffusion weighted (DW)-MRI imaging at the beginning, and on day 15+/-7 post treatment will be performed. Additionally, dual contrast enhanced CT (DECT) will be performed according to routine clinical evaluation time points before drug administration and at 8 weeks after drug administration. Disease will be monitored with serial CT scans of the chest abdomen and pelvis (CT-CAP) every eight weeks, until progression. The aim of the study is to identify novel predictive biomarkers of resistance and response to this targeted therapy in mCRC previously treated with oxaliplatin, fluoropyrimidines and irinotecan, using genetic, epigenetic, transcriptomics, proteomic and live tissue culture methods. These molecular analyses will be performed on metastatic tumour tissue samples taken firstly before commencement of regorafenib, and secondly on progression of disease, and thirdly from archival primary or metastatic tumour tissue. There is an additional biopsy at 8 weeks in patients with response or stable disease, as determined by Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with RAS mutant (MT) metastatic colorectal cancer (mCRC) who have been at least once treated with available therapies including fluoropyrimidine-based chemotherapy, oxaliplatin, irinotecan and an anti-angiogenic agent, except for patients who have not been treated with oxaliplatin due to previous documented peripheral neuropathy in an adjuvant setting or in those patients where disease has progressed within a short time from receiving adjuvant treatment (<12 months).
2. Eligible to receive regorafenib within the context of PROSPECT-R trial at the Royal Marsden Hospital

Exclusion criteria:

A patient who meets any of the exclusion criteria will NOT be eligible for randomization.

A patient must NOT

1. have had prior treatment with regorafenib or any other VEGF-targeting kinase inhibitor
2. have had previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer within 5 years prior to randomization EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (Noninvasive tumor), Tis (Carcinoma in situ) and T1 (Tumor invades lamina propria)].
3. Patients that are participating in another clinical trial involving an investigational medicinal product, unless it is more than 14 days after they have ceased the investigational medicinal product
4. Patients that are participating in another research study involving tumour tissue biopsies planned to take place during the time that the patient is participating in this study
5. Have had a major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to initiation of study treatment
6. If female and of childbearing potential, be engaged in breast feeding
7. Be unable to swallow oral tablets (crushing of study treatment tablets is not allowed)
8. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 month before the start of study medication (except for adequately treated catheter-related venous thrombosis occurring more than one month before the start of study medication)
9. Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
10. Ongoing infection > Grade 2 NCI Common Toxicity Criterial for Adverse Effects (CTCAE).
11. Uncontrolled hypertension (Systolic blood pressure > 140 mmHg or diastolic pressure > 90 mmHg) despite optimal medical management
12. Have congestive heart failure classified as New York Heart Association Class 2 or higher
13. Have had unstable angina (angina symptoms at rest) or new-onset angina < 3 months prior to screening
14. Have had a myocardial infarction < 6 months prior to initiation of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from the clinics and multi-disciplinary meetings, so long that they meet all the inclusion criteria and no exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2015-01; Primary Completion 2017-01 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
disease control rate (DCR), measured in months | 12 months
  DCR will be defined as complete response (CR)/partial response (PR)/ stable disease (SD) using RECIST v1.1. Chi2 or Fisher's exact tests will be employed to explore whether there is an association between low or high mutations and DCR. Logistic regression will be employed to produce odds ratios (ORs) and 95% confidence intervals (CIs).

SECONDARY OUTCOMES:
progression free survival (PFS), measured in months | 12 months
  PFS will be measured from start of treatment to date of progression or death from any cause.Logistic regression will be employed to produce odds ratios (ORs) and 95% confidence intervals (CIs). The PFS will be estimated using the Kaplan-Meier method and survival curves will be generated for each group. The log-rank test will be used to compare the survival curves and a Cox proportional hazards model will be fitted to obtain hazard ratios (HRs) and 95% CIs. The proportional hazards assumption will be tested with the use of Schoenfeld residuals
overall survival (OS), measured in months | 12 months
  OS will be defined as time from start of treatment to death of any cause. Logistic regression will be employed to produce odds ratios (ORs) and 95% confidence intervals (CIs). The OS will be estimated using the Kaplan-Meier method and survival curves will be generated for each group. The log-rank test will be used to compare the survival curves and a Cox proportional hazards model will be fitted to obtain hazard ratios (HRs) and 95% CIs. The proportional hazards assumption will be tested with the use of Schoenfeld residuals
Median values of volume transfer constant (Ktrans) and enhancing fraction (EF) and their product KEF (product of summarised median values of Ktrans x EF/100) will be compared at baseline and on day 15 | 15 days
  Dynamic contrast enhance magnetic resonance imaging (DCE-MRI) will be performed pre-treatment and at day 15. KEF changes of more than 70% between the two time points will be considered significant and patients will be thus stratified in two groups, i.e. A) drop in KEF of >70% and B) less than 70% drop in KEF.

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHS Foundation Trust London and Surrey, Carshalton, Surrey, United Kingdom

REFERENCES:
- [Derived] Rata M, Khan K, Collins DJ, Koh DM, Tunariu N, Bali MA, d'Arcy J, Winfield JM, Picchia S, Valeri N, Chau I, Cunningham D, Fassan M, Leach MO, Orton MR. DCE-MRI is more sensitive than IVIM-DWI for assessing anti-angiogenic treatment-induced changes in colorectal liver metastases. Cancer Imaging. 2021 Dec 19;21(1):67. doi: 10.1186/s40644-021-00436-0. PMID 34924031